CLINICAL TRIAL: NCT01093950
Title: White Light Scanning to Aid Body Contouring: A Pilot Project
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: Novaptus Systems Incorporated (Industry)
Responsible Party: Principal Investigator, David Gilbert, Principal Investigator, Eastern Virginia Medical School
Other Study IDs: 05-09-FB-0235
Record Dates: First submitted 2010-03-09; First posted 2010-03-26 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Lipodystrophy; Body Dysmorphic Disorders
Keywords: anthropometric; white light scanner; extraction profiles; Body lipodystrophy
MeSH Terms: conditions — Lipodystrophy; Body Dysmorphic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PROSPECTIVE BODY CONTOURING SUBJECTS: It is anticipated that the participants will undergo body contouring procedures including lipoplasty [internal fat suction removal], abdominoplasty [surgical removal of lower abdominal skin and fat], breast reduction [surgical removal of breast skin, fat, and breast tissue to reduce breast size], breast augmentation [surgical breast enlargement], thigh lift [surgical removal of upper thigh tissue], and brachioplasty [surgical removal of upper arm tissue].
  These procedures will be evaluated by pre- and post-operative digital scans, analog measurements, and clinical examinations and photographs.

SUMMARY:
A white light scanner can more accurately measure body contouring subjects than standard anthropomorphic methods.

DETAILED DESCRIPTION:
A 3-D digital body camera that employs non-intrusive white light phase profilometry and 24 coordinated charge-coupled cameras scans and produces a "point cloud" image of the subject. The result of the two-minute scan process is an accurate three-dimensional body model of the subject, consisting of over 1.2 million surface points. The point cloud is compressed to provide programmable measurement extraction profiles (MEP's) that automatically extracts linear and circumferential measurements. Subjects are scanned and anthropometrically measured pre-operatively, and at 3, 6 and 9 months post-op.

ELIGIBILITY:
Inclusion Criteria:

* All healthy preoperative body contouring subjects between 18-65 years old are potentially included in this study.

Exclusion Criteria:

* Pregnant, nursing,or have a history of epilepsy.
* Individuals under 18 years old;
* Problems reading or understanding spoken instructions;
* Are in jail or in a "locked ward";
* Are a student or an employee of EVMS; or
* Are chemically-dependent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy, prospective, surgical candidates for body contouring surgery, including: lipoplasty, abdominoplasty, breast reduction, breast augmentation, thigh lift,and brachioplasty are being asked to participate in this research project.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2005-01; Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
To study whether the scanner was faster and more accurate than anthropometric measurements. | 9 months
  The scanner and anthropometric measurements will be compared for accuracy and fidelity of collection. Anthropometric tape measurements will be compared to measurement extraction profiles provided by the scanner.Conclusions will be drawn based on the data collected.

CONTACTS AND LOCATIONS:
Overall Officials: David A Gilbert, MD, Principal Investigator — Eastern Virginia Medical School
Locations (1):
- The Hague Center, Norfolk, Virginia, United States